CLINICAL TRIAL: NCT03226925
Title: Added Value of Mechanically-assisted Ventilation in the Treatment of Moving Tumours (Thoracic/Upper Abdomen) With Photon and Proton Therapies.
Brief Title: Mechanically-assisted Ventilation in the Treatment of Moving Tumours With Photon and Proton Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/23MAI/294
Record Dates: First submitted 2017-06-27; First posted 2017-07-24 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Thoracic Neoplasm; Liver Cancer; Ventilator Lung; Radiotherapy; Complications
Keywords: thoracic tumors; motion management; radiotherapy; ventilator
MeSH Terms: conditions — Thoracic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: One group of patients with healthy volunteers and two groups with lung/upper abdomen cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers on ventilation (Experimental): Dynamic MRI acquisition will be performed at two different time points with 10 healthy volunteers under non-invasive mechanically-assisted ventilation with a respirator. Different modes will be compared (spontaneous, physiologic, shallow, slow and jet ventilation).
  Interventions: Diagnostic Test: Non-invasive mechanically-assisted ventilation; Diagnostic Test: Dynamic MRI acquisition
- Cancer patients on ventilation (Experimental): Dynamic MRI acquisition will be performed at two different time points with 10 patients (intended for a radiation treatment of their thoracic or upper abdominal tumours) under non-invasive mechanically-assisted ventilation with a respirator. Different modes will be compared (spontaneous, physiologic, shallow, slow and jet ventilation).
  Interventions: Diagnostic Test: Non-invasive mechanically-assisted ventilation; Diagnostic Test: Dynamic MRI acquisition
- Planning with patients on ventilation (Experimental): Planning 4D-CT will be performed with 10 patients (intended for a radiation treatment of their thoracic or upper abdominal tumours) under non-invasive mechanically-assisted ventilation with a respirator. Different ventilation modes will be compared (spontaneous, physiologic, shallow, slow and jet ventilation).
  Interventions: Diagnostic Test: Non-invasive mechanically-assisted ventilation; Diagnostic Test: Planning 4D-CT

INTERVENTIONS:
Diagnostic Test: Non-invasive mechanically-assisted ventilation — Mechanically ventilation will be done through facial masks connected to a respirator. Volunteers/patients are fully conscious during the ventilation.
Diagnostic Test: Dynamic MRI acquisition — Dynamic MRI acquisition are specific dynamic sequences intended to visualise the motion of internal structures (anatomical structures or tumour) under non-invasive mechanically-assisted ventilation
  Arms: Cancer patients on ventilation; Healthy volunteers on ventilation
Diagnostic Test: Planning 4D-CT — In order to perform in-silico planning, 4D-CT will be acquired on patients under non-invasive mechanically-assisted ventilation
  Arms: Planning with patients on ventilation

SUMMARY:
Mechanical ventilation can be used to impose a completely regular pattern of breathing frequency and inflation volume on the patient for as long as required. This would considerably improve the reproducibility of the internal motion parameters, and thus facilitate the implementation of respiratory-synchronized techniques such as gating, tracking and four-digital optimization.

DETAILED DESCRIPTION:
This will be a three-phase analysis :

First, different ventilation modes will be tested and compared on healthy volunteers. This phase will be analysed with a ventilator and with dynamic MRI in order to measure the movement of anatomical structures in each ventilation mode (intra-fraction analysis). Further, we will repeat these exams in order to compare them with the first ones, in order to analyse the reproducibility and baseline shifts (inter-fraction analysis).

Here are the different ventilation modes

* spontaneous breathing
* physiologic ventilation mode :
* shallow ventilation mode
* slow ventilation mode
* Jet Ventilation mode

Second phase will be done with patients that are intended to have a radiation treatment for thoracic or upper abdominal tumors. All the previous ventilation modes will be analysed during repeated MRI, again in order to perform intra- and inter-fraction analysis of the tumor motion.

Third phase also concerned patients intended to have a radiation treatment. It will be an in-silico-planning analysis in order to quantify dosimetric outcomes of these ventilation modes.

ELIGIBILITY:
Inclusion Criteria:

* No comorbidity for healthy volunteers
* Cancer patients with either lung or upper abdomen (liver/pancreas) tumours treated with radiation therapy.

Exclusion Criteria:

* severe lung disease or emphysema
* previous history of pneumothorax
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Measure in millimeters of the internal motion during non-invasive mechanically assisted ventilation, based on MRI images | within 12 months
  This analysis will be based on dynamic MRI analysis made with healthy volunteers and also patients on non-invasive mechanically assisted ventilation. A well defined anatomical structure will be selected for the healthy volunteers while the tumor will be tracked in patients.

SECONDARY OUTCOMES:
Tolerance assessment | within 12 months
  During all these acquisitions, the tolerance to the non-invasive mechanically assisted ventilation will be assessed by all the participants through a 5-steps scale.
Internal motion reproducibility with non-invasive mechanically assisted ventilation. | Within 12 months
  This analysis will be done by comparing the motion of the internal structures/tumors at two different time points (MRI acquisition at two different time points). All these acquisitions will obviously be done in the same conditions on non-invasive mechanically assisted ventilation. Motion reproducibility will be analysed by comparing the baseline positions of anatomical structures/tumors on MRI images and the measures in millimeters of motion of the same anatomical structures/tumors.
Dosimetric comparison | within 12 months
  This dosimetric comparison will be done in order to assess the impact of non-invasive mechanically-assisted ventilation on dose planning and delivery. Difference in dose (in Gy) to organ at risks will specially be compared through the DVH (dose-volume histogram) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Geets, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Not decided at this moment